CLINICAL TRIAL: NCT03024931
Title: In Vivo Cellular and Physiological Response to Severe Burns Injuries
Brief Title: Metabolic Rate in Burns
Acronym: MrBurn
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Marcela P. Vizcaychipi, Consultant in Anaesthesia and Intensive Care Medicine Honorary Senior Clinical Lecturer Divisional Research Lead for Planned Care Surgery and Clinical Support, Chelsea and Westminster NHS Foundation Trust
Other Study IDs: qw
Record Dates: First submitted 2016-12-03; First posted 2017-01-19 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational study — No intervention

SUMMARY:
Severe burn patients are some of the most challenging critically ill patients with an extreme and continuous state of physiological stress. Patients tends to stay for a long period of time in intensive care unit to treat burns as well as dealing with complications that arises from the initial burns injury. Severe burns patients are notoriously known to loose weight. The word 'catabolism' is used medically. This theory of catabolism after a trauma was hypothesised in 1942 by Professor Curthberston and based on animal models. Since this date, despite medical technological advancement, there has been no research that confirms Professor Curthberston's theory. Investigators still do not know the exact mechanism by which the body changes from conserving energy to becoming catabolic. Furthermore, it remains unclear whether this change in catabolism is necessary to heal from burns injury.

This theoretical catabolism in burns patients is currently treated with nutritional supplement, use of medications including beta-blockers (suppresses heart rate and decreases blood pressure) and oxandrolone (formula which is similar to testosterone to build up muscles).

There are evidences to suggest that increase in weight loss worsens the outcome in burns injury. Both overfeeding or underfeeding patients can be detrimental. In this research, the exact changes in metabolic rate will be measured in the first 72 hours of the study using a calorimetry machine. In addition to the metabolic rate, the response to the heart, liver, kidneys and hormonal levels will be measured. By looking into these dynamic changes the investigator will be able to elucidate whether there is a real increase in metabolic rate. If there is, the investigator would also be able to tell the response of different organs and whether there are any hormones that could be responsible to inflicting the metabolic changes.

DETAILED DESCRIPTION:
1. Purpose of the study The purpose of this study is to gain a better understanding of the acute physiological and metabolic changes in severe burns injury. Unless clinicians understand the physiological effect in burns patients, clinicians are unable to develop new therapeutic interventions to halt the hyper metabolic changes in burns patient. This research will be looking into the acute resting basal metabolic changes in severe adult burns patients by using Quark RMR (indirect calorimetry). This equipment will allow the investigator to detect the metabolic switch in severe burns patients.

   In addition to the metabolic changes, 'Estimated cardiac output monitor' will be placed in conjunction with calculating the Fick principle. Heart rate and pulse oximeter will be monitored continuously. These adjuncts will allow the investigator to conclude whether hyper-metabolism is associated with hyper dynamic cardiovascular response to burns.

   Splanchnic circulation will be monitored using the LiMON indocyanine green test and intermittent intra-abdominal pressure will be monitored to assess whether there is a link between the metabolic rate and splanchnic circulation.
2. Objectives

   1. Primary Objective:

      Identifying the 'Ebb' phase and 'Flow' phase in acute burns injury
   2. Secondary Objectives:

1. To establish cardiovascular response to burns in the acute phase.

a. To establish cardiovascular response to hyper-catabolism, using ESCO (estimated cardiac output) 2. To asses the relationship between the splanchnic circulation and hyper-catabolism 3. To assess the feasibility of performing LiMON test and (Bispectral Index) BIS monitoring for future (Burns Intensive Care Unit) BICU patients 4. To optimize dietary recommendations for patients who are suffering from hyper-catabolic state

8. Study Design Summary: This is a prospective, observational study with intensive monitoring but no experimental intervention

a) Study Site and Duration: This study will be conducted on the adult Burns Intensive Care Unit (BICU), Chelsea and Westminster Foundation Trust, London, United Kingdom (UK). This is a tertiary referral hospital serving an area of North West London. The average annual admission for severe burns to BICU varies form 10 -15 patients. The study will be conducted from December 2015 to December 2019.

The BICU has facilities for ventilatory support, sedation and surgery of critically ill patients, with two-bed intensive care unit. Each bed is isolated with three senior trained intensive care nurses covering 24 hours. Critically ill burns participants will be monitored continuously by nurses and doctors with the use of non-invasive and invasive monitoring depending on their clinical needs as per standard clinical care.

f) Procedure

General History and Examination Upon enrolment, full history and examination will be performed, including detailed assessment of the respiratory system, extent and depth of burns, neurological examination, cardiovascular examination and excluding other potential trauma that the participants could have suffered from.

The results will be recorded on a designated record form. Participants will be re-assessed by a physician or nurse for the duration of continuous monitoring to independently assess blood pressure, heart rate, respiratory rate, oxygen saturation, cardiac output, Glasgow coma scale, sedation score, ventilator requirement, urine output, intra-abdominal pressure, splanchnic circulation, BIS, EEG, nitrogen balance, resting metabolic rate and temperature.

Daily follow up will include assessment for any complications of burns including sepsis, infection, inhalational injury, suspected Acute Respiratory Distress Syndrome, and suspected respiratory distress of uncertain aetiology. The decision to obtain imaging or other investigations to assess such complications will be made by the clinical team and the results will be archived as source documents.

In addition to above, venous blood sample will be taken to establish on the daily basis to monitor inflammatory markers, renal, liver, bone marrow function, electrolyte levels. Urinary nitrogen levels, plasma hormones including Thyroid stimulating hormone, T3, T4, cortisol levels, insulin, glucagon levels are taken daily. These tests will be completed by the clinical team.

Regular arterial line gas sample will be taken as guided by the clinical team.

Continuous monitoring Participants will undergo standard electrophysiological monitoring, cardiovascular monitoring including arterial line blood pressure monitoring, placement of estimated cardiac output monitoring and intra-abdominal pressure. These devices will be connected to a portable diagnostic recording system to aid the diagnosis of any physiological changes that occurs. The system comprises a central device, with a display screen, battery pack and memory card. The electrophysiological monitoring device will consists or three electrodes and wires which feeds into the central device ports. The electrodes will be attached to the participants' forehead; left central and right. The intra-abdominal pressure device consists of a transducer which is located in the urinary catheter. The wires which are connected to the transducers are then fed into the central device ports. The continuous estimated cardiac output monitoring devices consist of three cardiac electrodes, pulse oximetry device and wires, which are connected to the central device ports. The cardiac electrodes are placed to the participants' thorax and the pulse oximetry device is attached to the participants' digit either in the foot or hand.

The following sensors will be applied:

* Electrocardiogram: recording cardiac electrical activity to give three recorded and three derived traces
* Ventilator: recording airflow inhale and exhalation, flow rate, pressure, tidal volume, peep, type of ventilator mode.
* Pulse oximeter: recording arterial oxygen saturation and pulse rate The monitoring system will be applied to the participant once assent is obtained and after the initial management; drug administration, examination and other investigation are performed by the clinical team. The sensors will be applied with the goal of recording continuously for seventy two hours.

Intermittent monitoring Participant will undergo indirect calorimetry monitoring and LIMON test. Resting metabolic rate will be measured every 12 hourly for 72 hours using indirect calorimetry with Quark Resting Metabolic Rate (QUARK RMR) (COSMED, Rome, Italy). This device consist of canopy, ventilator tubing, heat and moisture exchange filter, air sample analyzing tubes, computer, gas analyzing chamber, calibration gas cylinder, air pump to calibrate the flow sensor, fuel cell, spirometry and Windows 8.0 computer which has COSMED Quark RMR software installed.

Participants are either ventilated or awake. Ventilated participants will have a gas analyzing tubing attached to the heat and moisture exchange filter which is fed unto the gas analyzing chamber. The flow meter is attached at the exhaust port at the back of the ventilator.

The measurement is taken until a steady resting state is achieved. This will normally vary from two minutes to 20 minutes. The results are automatically recorded onto the Quark RMR software. In order to achieve steady ventilation with little minimum bias flow the participants' Bispectral index is maintained between forty and sixty using medications such as propofol, fentanyl, midazolam or clonidine.

Liver and splanchnic circulation will be measured every 6 hourly using LIMON Liver Function Monitor (Liver Monitor, PULSION Medical Systems, Munich, Germany) The device consist of sensor, wires and monitor to display the instructions and results. The sensor is attached to the participants' earlobe, finger tips in the hand or foot. The indocyanine green dye (ICG) is injected into a vein. The results will be displayed onto the monitor.

If the recording is suboptimal due to loss of sensors or insufficient recording, it will be repeated.

All of the above equipments and monitoring system will be cleaned and disinfected according to the manufacturing advice and microbiology team. The standard operating procedures for the above equipments are described in the appendix.

Cessation of monitoring The recording system, or individual sensors will be removed immediately if it is required for clinical investigations or interventions. However, it is anticipated that most investigations and interventions will be able to proceed with the sensors in place. The device is expected to remain in place during patient re-positioning, airway management, delivery of oxygen, delivery of oral and IV medication and fluids and most imaging with the exception of magnetic resonance imaging.

BIS monitoring will be removed in the event of cardio-respiratory arrest. If study clinician is not present at the time of cardio-respiratory arrest, the monitor will detach without difficulty and will not impede or delay resuscitation efforts.

Date collection:

In addition to above data, the investigator be collecting the patients' demographics including apache II scoring, end organ function including liver function, renal function, haematological status, ventilator settings, arterial gas, urine output and temperature.

9. Data Analysis Analysis of recording Data will be exported from the monitoring devices after each recording and assessed for adequacy and quality.

All frontal lobe electroencephalogram will be analysed. If there is any EEG finding that are consist with seizures it will be reviewed by neurophysiologist. All resting metabolic rate will be plotted against the physiological parameters including splanchnic circulation, temperature and intra-abdominal pressure. The ECG will be reviewed to assess heart rate, rhythm and conduction. Invasive blood pressure monitoring device will assess the blood pressure. Estimated cardiac output monitoring will assess the cardiac output and the trend over the seventy two hours. Fick principle will be used to calculate the cardiac output using the data (CaO2 and CVO2) obtained from the Quark RMR.

Any stimulus, airway management, changes in the levels of sedation, return from theatres will be noted.

1. Statistical Consideration In the view of the complexity of data provided by continuous monitoring, statistical guidance will be sought at all stages of analysis from the "Statistician. For the primary end points, the investigator will draw a graph of time again resting metabolic rate. The precise choice of test will be determined once the distribution pattern of the data is known. Repeated measure analysis of variance will be used followed by regression analysis accounted for repeat measures.

   In comparing patient specific outcome measures (mortality, requirement for ventilation, development of complications such as sepsis), participants will be placed into ranked groups from most to least difference in trend change in resting metabolic rate and nonparametric analysis will be used to assess the relationship between mortality or morbidity and resting metabolic rate.
2. Sample Size Justification Primary determinant is expected number of eligible patients presenting in the duration of study.

Power calculation was completed for the primary outcome measures. In order to conclude to show that there is an increase in metabolic rate by 200 kcal per day with a power of 0.8, I will need 8 patients to be able to conclude that there increase in metabolic rate.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 16 years or over
* Informed, written consent from patient. If the participant is unable to give consent then assent will be considered.
* Burns more than 15%
* Acute presentation

Exclusion Criteria:

* Any concern from the clinical team that the application or ongoing presence of the monitoring device would interfere with optimal patient management.
* Allergy to adhesives used for monitor leads and belts.
* Participants below 16 years old
* Burns less than 5%
* Conditions that gives an inaccurate calorimetry results
* Participants needing oxygen concentration more than 60%
* Participants who have broncho-alveolar fistula
* Participants with chest drains
* Airway leak within the ventilated systems

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators plan to study 10 adult patients with severe burns participants within the first 72 hours of admission to the BICU. Participants will be recruited from the burns intensive care adult unit (BICU), CWFT, London, UK. Inclusion and exclusion criteria are below.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Monitor the change in resting metabolic rate over period of time after severe burns injury. | Continuous monitoring over 72 hours
  The resting metabolic rate will be measured using Quark Indirect Calorimetry Machine from Cosmed, Italy. The rested metabolic rate will be measured in kilo calories.

SECONDARY OUTCOMES:
Monitor the cardiac output using Fick principle in severe burns | The cardiac output will be measured using the fick principle.The cardiac output will be measured at 12th, 24th, 36th, 48th, 60th 72nd hour from the point of the injury. 10 patients will be recruited over a year.
  The cardiac output will be measured in mls.
Monitor the splanchnic circulation by measuring the indocyanine green clearance rate. | The splanchnic circulation will be measured at 12th, 24th, 36th, 48th, 60th 72nd hour from the point of the injury. 10 patients will be recruited over a year.
  splanchnic circulation will be measured by using Limon machine from Maquet. The plasma clearance rate of indocyanine green will be measured in % per ml.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Vizcaychipi, Principal Investigator — Chelsea and Westminster NHS trust
Locations (1):
- The Burn Intensive Care Unit (BICU), Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no, we do not plan to share participant data with other researchers.

REFERENCES:
- [Result] Herndon DN, Hart DW, Wolf SE, Chinkes DL, Wolfe RR. Reversal of catabolism by beta-blockade after severe burns. N Engl J Med. 2001 Oct 25;345(17):1223-9. doi: 10.1056/NEJMoa010342. PMID 11680441
- [Result] Huang YS, Yang ZC, Liu XS, Chen FM, He BB, Li A, Crowther RS. Serial experimental and clinical studies on the pathogenesis of multiple organ dysfunction syndrome (MODS) in severe burns. Burns. 1998 Dec;24(8):706-16. doi: 10.1016/s0305-4179(98)00123-5. PMID 9915670
- [Result] Jeschke MG, Gauglitz GG, Kulp GA, Finnerty CC, Williams FN, Kraft R, Suman OE, Mlcak RP, Herndon DN. Long-term persistance of the pathophysiologic response to severe burn injury. PLoS One. 2011;6(7):e21245. doi: 10.1371/journal.pone.0021245. Epub 2011 Jul 18. PMID 21789167
- [Result] Jeschke MG, Herndon DN, Wolf SE, DebRoy MA, Rai J, Lichtenbelt BJ, Barrow RE. Recombinant human growth hormone alters acute phase reactant proteins, cytokine expression, and liver morphology in burned rats. J Surg Res. 1999 May 15;83(2):122-9. doi: 10.1006/jsre.1999.5577. PMID 10329105
- [Result] Kasten KR, Makley AT, Kagan RJ. Update on the critical care management of severe burns. J Intensive Care Med. 2011 Jul-Aug;26(4):223-36. doi: 10.1177/0885066610390869. PMID 21764766
- [Result] CUTHBERTSON DP. Interrelationship of metabolic changes consequent to injury. Br Med Bull. 1954;10(1):33-7. doi: 10.1093/oxfordjournals.bmb.a069369. No abstract available. PMID 13126521
- [Result] CUTHBERTSON DP. Nutrition. Annu Rev Med. 1953;4:135-62. doi: 10.1146/annurev.me.04.020153.001031. No abstract available. PMID 13105270
- [Result] Bell JR, Clark AM, Cuthbertson DP. Experimental traumatic shock. J Physiol. 1938 May 14;92(4):361-70. doi: 10.1113/jphysiol.1938.sp003608. No abstract available. PMID 16994980
- [Result] Cathcart EP, Cuthbertson DP. The composition and distribution of the fatty substances of the human subject. J Physiol. 1931 Jul 6;72(3):349-60. doi: 10.1113/jphysiol.1931.sp002779. No abstract available. PMID 16994214